CLINICAL TRIAL: NCT07107828
Title: Effect of Rehabilitation on the Respiratory Signal in Patients With Chronic Obstrucitve Pulmonary Disease (COPD) and Exercise-Induced Desaturation
Brief Title: Effect of Rehabilitation on the Respiratory Signal in Patients With COPD and Exercise-Induced Desaturation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Switzerland University of Applied Sciences (Other)
Collaborators: University of Edinburgh (Other); National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: inRehaExO2_Respeck
Record Dates: First submitted 2025-07-16; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Rehabilitation; Exercise; Oxygen; Breathing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Respiratory Aspiration | interventions — Particulate Matter; Oxygen; Altitude

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normoxia (Sham Comparator): Sham air (ambient air) will be applied with the oxygen concentrator EverFloTM via nasal cannula
  Interventions: Other: Ambient air
- Hyperoxia (Active Comparator): Standardized supplemental oxygen (SSOT) will be applied with the oxygen concentrator EverFloTM via nasal cannula
  Interventions: Other: Oxygen
- Hypoxia (Experimental): This group will train at moderate altitude
  Interventions: Other: Altitude

INTERVENTIONS:
Other: Ambient air — Standard ambient air will be breathed during endurance training.
  Arms: Normoxia
Other: Oxygen — SSOT will be applied during endurance training
  Arms: Hyperoxia
Other: Altitude — Training will be performed at moderate altitude
  Arms: Hypoxia

SUMMARY:
The aim is to study the effect of SSOT during a 3-week in-patient pulmonary rehabilitation programme. Further aim is to analyse exercise endurance, distinguishing between those exercising whilst breathing air at 760m "normoxia", breathing air at 1600m "hypoxia", or breathing SSOT at 760m "hyperoxia" conditions, during in-patient pulmonary rehabilitation.

The objective of the main study is to provide long-awaited data concerning the use of SSOT during training. At present it is unclear whether patients with chronic lung diseases who reveal an SpO2 > 88% at rest, but desaturate during exercise, and, thus, may not qualify for long-term oxygen undergoing PR benefit from supplemental oxygen.

This sub-study will involve the subjects wearing the Respeck device and will focus on the effect of exercise on the respiratory signal measured by the Respeck.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years
* stable condition > 3 weeks (e.g. no exacerbations)
* resting SpO2 ≥ 88% and exercise induced hypoxemia defined by a fall in SpO2 by ≥ 4% and/or below 90% during a 6-minute walk test (6MWT)
* informed consent as documented by signature.

Exclusion Criteria:

* Severe daytime resting hypoxemia (SpO2 < 88%)
* long-term oxygen therapy
* unstable condition requiring adaptation of pharmacologic and other treatment modalities or requirement of intensive care or relevant severe concomitant disease
* inability to follow the procedures of the study, e.g. due to language problems psychological disorders, neurological or orthopedic problems with walking disability or inability to ride a bicycle
* women who are pregnant or breast feeding
* enrolment in another clinical trial with active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2025-07-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of respiratory rate (in terms of breaths/minute) | 3 weeks
  The longitudinal analysis of features extracted from the continuous Respeck respiratory flow/effort signals pre and post the 3-week in-house rehabilitation programme, and comparisons between the different groups.

SECONDARY OUTCOMES:
Comparison of respiratory rate (in terms of breaths/minute) | before and after 6-minute walking distance
  Analysis of the respiratory signal before and after 6-minute walking distance
Comparison of respiratory rate (in terms of breaths/minute) | before and after constant work rate exercise test
  Analysis of the respiratory signal before and after constant work rate exercise test
Comparison of respiratory rate (in terms of breaths/minute) | 3 weeks
  Analysis of the respiratory signal before and after exercise (6-minute walking distance and constant work rate exercise test), and comparing before and after rehabilitation.

CONTACTS AND LOCATIONS:
Locations (1):
- National center for cardiology and internal medicine, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: No
IPD will only be shared upon personal request to the corresponding author.